CLINICAL TRIAL: NCT03227029
Title: Randomized Phase I Study of the Infectivity, Safety, and Immunogenicity of a Single Dose of the Recombinant Live-Attenuated Respiratory Syncytial Virus (RSV) Vaccines RSV ΔNS2/Δ1313/I1314L or RSV 276 or Placebo, Delivered as Nose Drops to RSV-Seronegative Infants 6 to 24 Months of Age
Brief Title: Evaluating the Infectivity, Safety, and Immunogenicity of Recombinant Live-Attenuated RSV Vaccines RSV ΔNS2/Δ1313/I1314L or RSV 276 in RSV-Seronegative Infants 6 to 24 Months of Age
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IMPAACT 2018; 38405 (Registry Identifier: DAIDS-ES Registry Number); NCT03422237 (obsolete NCT alias)
Record Dates: First submitted 2017-07-20; First posted 2017-07-24 (Actual); Results first posted 2021-01-08 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Respiratory Syncytial Virus Infections
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- RSV ΔNS2/Δ1313/I1314L vaccine (Experimental): Participants received a single dose of the RSV ΔNS2/Δ1313/I1314L vaccine at study entry (Day 0).
  Interventions: Biological: RSV ΔNS2/Δ1313/I1314L
- RSV 276 vaccine (Experimental): Participants received a single dose of the RSV 276 vaccine at study entry (Day 0).
  Interventions: Biological: RSV 276
- Placebo (Placebo Comparator): Participants received a single dose of placebo at study entry (Day 0).
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: RSV ΔNS2/Δ1313/I1314L — 10^6 plaque-forming units (PFU); administered as nose drops
  Arms: RSV ΔNS2/Δ1313/I1314L vaccine
Biological: RSV 276 — 10^5 PFU; administered as nose drops
  Arms: RSV 276 vaccine
Biological: Placebo — Isotonic diluent, administered as nose drops
  Arms: Placebo

SUMMARY:
The purpose of this study was to evaluate the infectivity, safety, and immunogenicity of the recombinant live-attenuated respiratory syncytial virus (RSV) vaccines RSV ΔNS2/Δ1313/I1314L or RSV 276 when delivered as nose drops to RSV-seronegative infants 6 to 24 months of age.

This study was a companion study to Center for Immunization Research (CIR) 321.

DETAILED DESCRIPTION:
Human respiratory syncytial virus (RSV) is the most common viral cause of serious acute lower respiratory illness (LRI) in infants and children under 5 years of age worldwide. This study evaluated the infectivity, safety, and immunogenicity of two recombinant live-attenuated RSV vaccines: RSV ΔNS2/Δ1313/I1314L and RSV 276. The vaccines were delivered as nose drops to RSV-seronegative infants 6 to 24 months of age.

Participants were randomly assigned to receive a single dose of the RSV ΔNS2/Δ1313/I1314L vaccine, the RSV 276 vaccine, or placebo at study entry (Day 0).

Participants could be enrolled in the study outside of RSV season, i.e., between April 1 and October 14 for most sites or-for sites with local RSV seasons that start earlier-as specified on a site-by-site basis in the manual of procedures. Participants remained on study until they completed the post-RSV season visit between April 1 and April 30 in the calendar year following enrollment. Participants' total study duration was between 6 and 13 months, depending on when they enrolled in the study. Participants attended several study visits throughout the study, which included physical examinations, blood collection, nasal washes, and/or nasal adsorption (nasosorption) specimen collection. Participants' parents or guardians were contacted by study staff at various times during the study to monitor participants' health.

ELIGIBILITY:
Inclusion Criteria:

* In good health based on review of the medical record, history, and physical examination, without evidence of chronic disease.
* Parent/guardian willing and able to provide written informed consent as described in the protocol.
* Seronegative for RSV antibody, defined as a serum RSV-neutralizing antibody titer less than 1:40 at screening from a sample collected no more than 42 days prior to inoculation.
* Growing normally for age (i.e., not downwardly crossing two major centiles on a standard growth chart) in the six months prior to enrollment AND

  * If less than 1 year of age: current height and weight above the 5th percentile
  * If 1 year of age or older: current height and weight above the 3rd percentile for age.
* Received routine immunizations appropriate for age (as per national Center for Disease Control Advisory Committee on Immunization Practices).
* Expected to be available for the duration of the study.
* If born to an HIV-infected woman, participant must not have been breastfed and must have documentation of 2 negative HIV nucleic acid (RNA or DNA) test results from samples collected on different dates with both collected when greater than or equal to 4 weeks of age and at least one collected when greater than or equal to 16 weeks of age, and no positive HIV nucleic acid (RNA or DNA) test; or 2 negative HIV antibody tests, both from samples collected at greater than or equal to 24 weeks of age.

Exclusion Criteria:

* Known or suspected HIV infection or impairment of immunological functions.
* Receipt of immunosuppressive therapy, including any systemic, including either nasal or inhaled, corticosteroids within 28 days of enrollment. Note: Cutaneous (topical) steroid treatment is not an exclusion.
* Any receipt of bone marrow/solid organ transplant.
* Major congenital malformations (such as congenital cleft palate) or cytogenetic abnormalities.
* Previous receipt of a licensed or investigational RSV vaccine (or placebo in any International Maternal Pediatric Adolescent AIDS Clinical Trials Network RSV study) or previous receipt of or planned administration of any anti-RSV product (such as ribavirin or RSV IG or RSV mAb).
* Any previous anaphylactic reaction.
* Any previous vaccine-associated adverse reaction that was Grade 3 or above. Note: if grading is not possible, determine if the reaction was considered severe or life threatening; if so, it is exclusionary.
* Any known hypersensitivity to any study product component.
* Heart disease. Note: Participants with cardiac abnormalities documented to be clinically insignificant and requiring no treatment may be enrolled.
* Lung disease, including any history of reactive airway disease or medically diagnosed wheezing.
* Member of a household that contained, or would contain, an infant who is less than 6 months of age at the enrollment date through Day 28.
* Member of a household that contained another child/other children who was/were, or was/were scheduled to be, enrolled in IMPAACT 2018 AND the date of enrollment to IMPAACT 2018 would not be concurrent with the other participant(s) living in the household (i.e., all eligible children from the same household must be enrolled on the same date).
* Member of a household that contained another child who was, or was scheduled to be, enrolled in another study evaluating an intranasal live-attenuated RSV vaccine, AND there has been or would be an overlap in residency during that other child's participation in the study's Acute Phase (Days 0 to 28).
* Member of a household that contained an immunocompromised individual, including, but not limited to:

  * a person who was greater than or equal to 6 years of age with HIV-related immunodeficiency, defined as having a most recent CD4 T lymphocyte cell count less than 300 cells/mm^3. CD4 T lymphocyte count must have been measured within 6 months prior to enrollment for individuals with detectable virus or within 12 months prior to enrollment for individuals with undetectable virus, or
  * a person age 1 year up to less than 6 years with HIV-related immunodeficiency, defined as having a most recent CD4 T lymphocyte cell percentage less than 25 or CD4 T lymphocyte count less than 750 cells/mm^3 (if both values are available, use the lower of the two). CD4 T lymphocyte parameter must have been measured within the 6 months prior to enrollment; or
  * a person age less than 1 year with HIV-related immunodeficiency, defined as having a most recent CD4 T lymphocyte cell percentage less than 30 or CD4 T lymphocyte count less than 1000 cells/mm^3 (if both values are available, use the lower of the two). CD4 T lymphocyte parameter must have been measured within the 6 months prior to enrollment; or
  * a person who had received chemotherapy within the 12 months prior to enrollment; or
  * a person receiving immunosuppressant agents; or
  * a person living with a solid organ or bone marrow transplant. Documenting the verbal report of CD4 T cell lymphocyte count was sufficient if the parent/guardian was confident of history. Individually identifiable information (e.g., name) pertaining to members of the household were not collected or recorded. Confirmatory laboratory tests for members of the household were not ordered or collected.
* Attended a daycare facility and shared a room with infants less than 6 months of age, and parent/guardian was unable or unwilling to suspend daycare for 28 days following inoculation.
* Any of the following events at the time of enrollment:

  * fever (rectal temperature of greater than or equal to 100.4°F (38°C)), or
  * upper respiratory signs or symptoms (rhinorrhea, cough, or pharyngitis) or
  * nasal congestion significant enough to interfere with successful inoculation, or
  * otitis media.
* Receipt of the following prior to enrollment:

  * any inactivated vaccine or live-attenuated rotavirus vaccine within the 14 days prior, or
  * any live vaccine, other than rotavirus vaccine, within the 28 days prior, or
  * another investigational vaccine or investigational drug within 28 days prior
* Scheduled administration of the following after planned inoculation:

  * inactivated vaccine or live-attenuated rotavirus vaccine within the 14 days after, or
  * any live vaccine other than rotavirus in the 28 days after, or
  * another investigational vaccine or investigational drug in the 56 days after
* Receipt of immunoglobulin, any antibody products, or any blood products within the past 6 months prior to enrollment.
* Receipt of any of the following medications within 3 days prior to study enrollment:

  * systemic antibacterial, antiviral, antifungal, anti-parasitic, or antituberculous agents, whether for treatment or prophylaxis, or
  * intranasal medications, or
  * other prescription medication except as listed below. Permitted concomitant medications (prescription or non-prescription) include nutritional supplements, medications for gastroesophageal reflux, eye drops, and topical medications, including (but not limited to) cutaneous (topical) steroids, topical antibiotics, and topical antifungal agents.
* Receipt of salicylate (aspirin) or salicylate-containing products within the 28 days prior to enrollment.
* Born at less than 34 weeks gestation.
* Born at less than 37 weeks gestation and less than 1 year of age at the time of enrollment.
* Current suspected or documented developmental disorder, delay, or other developmental problem.
* Any previous receipt of supplemental oxygen therapy in a home setting.

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 65 (Actual)
Dates: Start 2017-09-22 (Actual); Primary Completion 2019-12-19 (Actual); Study Completion 2020-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Coleen Cunningham, MD, Study Chair — Children's Health Center, DUMC
Locations (12):
- United States (12):
  - University of California, UC San Diego CRS- Mother-Child-Adolescent HIV Program, La Jolla, California
  - Usc La Nichd Crs, Los Angeles, California
  - David Geffen School of Medicine at UCLA NICHD CRS, Los Angeles, California
  - Univ. of Colorado Denver NICHD CRS, Aurora, Colorado
  - Rush Univ. Cook County Hosp. Chicago NICHD CRS, Chicago, Illinois
  - Lurie Children's Hospital of Chicago (LCH) CRS, Chicago, Illinois
  - Johns Hopkins University Center for Immunization Research, Baltimore, Maryland
  - Boston Medical Center Ped. HIV Program NICHD CRS, Boston, Massachusetts
  - SUNY Stony Brook NICHD CRS, Stony Brook, New York
  - Jacobi Med. Ctr. Bronx NICHD CRS, The Bronx, New York
  - St. Jude Children's Research Hospital CRS, Memphis, Tennessee
  - Texas Children's Hospital CRS, Houston, Texas

REFERENCES:
- [Derived] Cunningham CK, Karron RA, Muresan P, Kelly MS, McFarland EJ, Perlowski C, Libous J, Oliva J, Jean-Philippe P, Moye J, Schappell E, Barr E, Rexroad V, Johnston B, Chadwick EG, Cielo M, Paul M, Deville JG, Aziz M, Yang L, Luongo C, Collins PL, Buchholz UJ; International Maternal Pediatric Adolescent AIDS Clinical Trials (IMPAACT) 2018 Study Team. Evaluation of Recombinant Live-Attenuated Respiratory Syncytial Virus (RSV) Vaccines RSV/DeltaNS2/Delta1313/I1314L and RSV/276 in RSV-Seronegative Children. J Infect Dis. 2022 Dec 13;226(12):2069-2078. doi: 10.1093/infdis/jiac253. PMID 35732186
- See also: Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events (Corrected Version 2.1 - July 2017) — http://rsc.niaid.nih.gov/sites/default/files/daidsgradingcorrectedv21.pdf
- See also: Manual for Expedited Reporting of Adverse Events to DAIDS (DAIDS EAE Manual), Version 2.0, January 2010 — http://rsc.niaid.nih.gov/clinical-research-sites/manual-expedited-reporting-adverse-events-daids

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period was from September 2017 to October 2019. Participants were recruited from 12 medical clinics all in the United States.
Period: Overall Study
Arm/Group | RSV ΔNS2/Δ1313/I1314L Vaccine | RSV 276 Vaccine | Placebo
Started | 26 | 26 | 13
Received Inoculation | 26 | 25 | 12
Completed | 22 | 22 | 9
Not Completed | 4 | 4 | 4
Not completed — Child Wheezed (no treatment) | 0 | 1 | 0
Not completed — No post RSV season visit due to COVID | 3 | 3 | 2
Not completed — Not able to get to clinic | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Unable to receive treatment in time (no treatment) | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline analysis population was participants who received inoculation and were followed on study past Day 0.
Groups:
- Total: Total of all reporting groups
Arm/Group | RSV ΔNS2/Δ1313/I1314L Vaccine | RSV 276 Vaccine | Placebo | Total
Number analyzed (Participants) | 25 | 25 | 12 | 62
Age, Continuous [Median (Inter-Quartile Range); unit: months] | 13 [7 to 14] | 14 [10 to 16] | 9 [7.5 to 14.5] | 12.5 [8 to 15]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 7 | 9 | 29
  Male | 12 | 18 | 3 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 9 | 3 | 21
  Not Hispanic or Latino | 15 | 16 | 9 | 40
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 7 | 7 | 6 | 20
  White | 15 | 14 | 6 | 35
  More than one race | 2 | 2 | 0 | 4
  Unknown or Not Reported | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 12 | 62
Serum RSV-neutralizing antibody titers [Median (Inter-Quartile Range); unit: Log 2 titers] | 2.3 [2.3 to 3.3] | 2.3 [2.3 to 2.3] | 2.3 [2.3 to 2.9] | 2.3 [2.3 to 2.3]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Solicited Adverse Events (AEs) by Grade
Description: Solicited adverse events included fever; otitis media; upper respiratory illness (URI); lower respiratory illness (LRI) and cough (without LRI). The number of participants who experienced solicited adverse events was presented. A participant was only counted once in each solicited AE category, and that is in the line corresponding to the highest grade adverse event they had in that category. These events were graded (Grade 1-mild to Grade 4-life-threatening) following protocol-defined grading system outlined in Table 5 and Table 6 in the protocol document.
Time Frame: Measured from Day 0 through Day 28
Population: Study participants who received inoculation and were followed on study past Day 0 were included.
Measure: Count of Participants; unit: Participants
Arm/Group | RSV ΔNS2/Δ1313/I1314L Vaccine | RSV 276 Vaccine | Placebo
Number analyzed (Participants) | 25 | 25 | 12
Participants
  Fever: Did not have this AE | 21 | 22 | 11
  Fever: Grade 1 | 1 | 0 | 0
  Fever: Grade 2 | 1 | 2 | 1
  Fever: Grade 3 | 2 | 1 | 0
  Fever: Grade 4 | 0 | 0 | 0
  Otitis Media: Did not have this AE | 24 | 23 | 12
  Otitis Media: Grade 1 | 0 | 0 | 0
  Otitis Media: Grade 2 | 1 | 2 | 0
  Otitis Media: Grade 3 | 0 | 0 | 0
  Otitis Media: Grade 4 | 0 | 0 | 0
  Upper Respiratory Illness (URI): Did not have this AE | 9 | 7 | 7
  Upper Respiratory Illness (URI): Grade 1 | 16 | 16 | 5
  Upper Respiratory Illness (URI): Grade 2 | 0 | 2 | 0
  Upper Respiratory Illness (URI): Grade 3 | 0 | 0 | 0
  Upper Respiratory Illness (URI): Grade 4 | 0 | 0 | 0
  Lower Respiratory Illness (LRI) with RSV shedding: Did not have this AE | 25 | 25 | 12
  Lower Respiratory Illness (LRI) with RSV shedding: Grade 1 | 0 | 0 | 0
  Lower Respiratory Illness (LRI) with RSV shedding: Grade 2 | 0 | 0 | 0
  Lower Respiratory Illness (LRI) with RSV shedding: Grade 3 | 0 | 0 | 0
  Lower Respiratory Illness (LRI) with RSV shedding: Grade 4 | 0 | 0 | 0
  LRI in the absence of RSV shedding: Did not have this AE | 25 | 25 | 12
  LRI in the absence of RSV shedding: Grade 1 | 0 | 0 | 0
  LRI in the absence of RSV shedding: Grade 2 | 0 | 0 | 0
  LRI in the absence of RSV shedding: Grade 3 | 0 | 0 | 0
  LRI in the absence of RSV shedding: Grade 4 | 0 | 0 | 0
  Cough, without LRI: Did not have this AE | 22 | 13 | 10
  Cough, without LRI: Grade 1 | 3 | 11 | 1
  Cough, without LRI: Grade 2 | 0 | 1 | 1
  Cough, without LRI: Grade 3 | 0 | 0 | 0
  Cough, without LRI: Grade 4 | 0 | 0 | 0
Statistical Analysis 1: Comparison: RSV ΔNS2/Δ1313/I1314L Vaccine; Test type: Other; % vaccine recipients with solicited AEs = 64, 90% CI 2-sided [46 to 80] — Proportions of study participants were calculated and presented with 90% exact confidence intervals. This highlights that we are 95% sure that the true proportion is not higher that the upper limit of the confidence interval
Statistical Analysis 2: Comparison: RSV 276 Vaccine; Test type: Other; % vaccine recipients with solicited AEs = 84, 90% CI 2-sided [67 to 94]
Statistical Analysis 3: Comparison: Placebo; Test type: Other; % placebo recipients with solicited AEs = 58, 90% CI 2-sided [32 to 82]

2. Primary Outcome: Number of Participants With Unsolicited AEs
Description: Unsolicited adverse events were other events, not included in the solicited AEs. The number of participants who experienced solicited adverse events was presented. A participant was only counted once in each unsolicited AE category, and that is in the line corresponding to the highest grade adverse event they had in that category. AE grading (Grade 1- mild to Grade 4-life-threatening) was done by Division of AIDS (DAIDS) AE Grading table v2.0 (see References).
Time Frame: Measured from Day 0 through Day 28
Population: Study participants who received inoculation and were followed on study past Day 0 were included.
Measure: Count of Participants; unit: Participants
Arm/Group | RSV ΔNS2/Δ1313/I1314L Vaccine | RSV 276 Vaccine | Placebo
Number analyzed (Participants) | 25 | 25 | 12
Participants | 9 | 13 | 5
Statistical Analysis 1: Comparison: RSV ΔNS2/Δ1313/I1314L Vaccine; Test type: Other; % vaccine recipients with usolicited AEs = 36, 90% CI 2-sided [20 to 54]
Statistical Analysis 2: Comparison: RSV 276 Vaccine; Test type: Other; % vaccine recipients with usolicited AEs = 52, 90% CI 2-sided [34 to 69]
Statistical Analysis 3: Comparison: Placebo; Test type: Other; % placebo recipients with usolicited AEs = 42, 90% CI 2-sided [18 to 68]

3. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: A Serious Adverse Event (SAE) is an AE, whether considered related to the study product or not, that:
  * Results in death during the period of protocol-defined surveillance;
  * Is life threatening: defined as an event in which the patient was at immediate risk of death at the time of the event; it does not refer to an event that hypothetically might have caused death were it more severe;
  * Requires inpatient hospitalization (or prolongation of existing hospitalization): defined as at least an overnight stay in the hospital or emergency ward for treatment that would have been inappropriate if administered in the outpatient setting;
  * Results in a persistent or significant disability/incapacity;
  * Is a congenital anomaly or birth defect, OR
  * Is an important medical event that may not be immediately life threatening or result in death or hospitalization but may jeopardize the patient or may require intervention to prevent one of the outcomes listed above.
Time Frame: Measured from Day 0 through Day 56
Population: Study participants who received inoculation and were followed on study past Day 0 were included.
Measure: Count of Participants; unit: Participants
Arm/Group | RSV ΔNS2/Δ1313/I1314L Vaccine | RSV 276 Vaccine | Placebo
Number analyzed (Participants) | 25 | 25 | 12
Participants | 0 | 0 | 0

4. Primary Outcome: Number of Participants Infected With RSV Vaccine Virus
Description: Defined as 1) vaccine virus identified in a nasal wash from Study Day 0-28 (a binary outcome based on nasal washes); and/or 2) greater than or equal to 4-fold rise in RSV serum neutralizing antibody titer and/or serum enzyme-linked immunosorbent assay (ELISA) titer to the RSV F protein from study entry to Study Day 56
Time Frame: Measured at Days 0, 3, 5, 7, 10, 12, 14, 17, and 28 for nasal washes, and at Days 0, 56 for serum RSV-neutralizing antibodies
Population: Study participants who received inoculation and were followed on study past Day 0 were included. One child from a set of twins was randomly selected and excluded from the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | RSV ΔNS2/Δ1313/I1314L Vaccine | RSV 276 Vaccine | Placebo
Number analyzed (Participants) | 25 | 24 | 12
Participants | 22 | 23 | 0
Statistical Analysis 1: Comparison: RSV ΔNS2/Δ1313/I1314L Vaccine; Test type: Other; % recipients infected with vaccine virus = 88, 90% CI 2-sided [72 to 97]
Statistical Analysis 2: Comparison: RSV 276 Vaccine; Test type: Other; % recipients infected with vaccine virus = 96, 90% CI 2-sided [82 to 100]
Statistical Analysis 3: Comparison: Placebo; Test type: Other; % recipients infected with vaccine virus = 0, 90% CI 2-sided [0 to 22]

5. Primary Outcome: Peak Titer of Vaccine Virus Shed
Description: This is the highest value per participant of the titer of vaccine virus shed. It was measured by culture. Only participants who met the definition of infection with vaccine virus were included.
Time Frame: Measured at Days 0, 3, 5, 7, 10, 12, 14, 17, and 28
Population: Only participants who met the definition of infection with vaccine virus were included.
Measure: Median (Inter-Quartile Range); unit: log 10 PFU/mL
Arm/Group | RSV ΔNS2/Δ1313/I1314L Vaccine | RSV 276 Vaccine | Placebo
Number analyzed (Participants) | 22 | 23 | 0
log 10 PFU/mL | 3.1 [1.8 to 3.8] | 3.2 [2.8 to 4.0] |

6. Primary Outcome: Duration of Virus Shedding in Nasal Washes
Description: Determined separately by a) culture and b) reverse transcription polymerase chain reaction (RT-PCR)
Time Frame: Measured at Days 0, 3, 5, 7, 10, 12, 14, 17, and 28. Last day positive is reported.
Population: Only participants who met the definition of infection with vaccine virus were included.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | RSV ΔNS2/Δ1313/I1314L Vaccine | RSV 276 Vaccine | Placebo
Number analyzed (Participants) | 22 | 23 | 0
days
  Culture positive | 10 [8 to 12] | 10 [7 to 12] |
  RT-PCR positive | 13 [12 to 16] | 14 [11 to 17] |

7. Primary Outcome: Number of Participants With a Greater Than or Equal to 4-fold Rise in Serum RSV-neutralizing Antibody Titers
Description: Antibody responses were defined as a greater than or equal to 4-fold increase in titer in paired specimens, between pre-inoculation and post-inoculation time points.
Time Frame: Measured at Day 0 and Day 56
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | RSV ΔNS2/Δ1313/I1314L Vaccine | RSV 276 Vaccine | Placebo
Number analyzed (Participants) | 25 | 24 | 12
Participants | 15 | 22 | 0
Statistical Analysis 1: Comparison: RSV ΔNS2/Δ1313/I1314L Vaccine; Test type: Other; % with >=4 fold rise in RSV-PRNT = 60, 90% CI 2-sided [42 to 76]
Statistical Analysis 2: Comparison: RSV 276 Vaccine; Test type: Other; % with >=4 fold rise in RSV-PRNT = 92, 90% CI 2-sided [76 to 98]
Statistical Analysis 3: Comparison: Placebo; Test type: Other; % with >=4 fold rise in RSV-PRNT = 0, 90% CI 2-sided [0 to 22]
Statistical Analysis 4: Comparison: RSV ΔNS2/Δ1313/I1314L Vaccine vs Placebo; Test type: Superiority; p < 0.01, Fisher Exact — Due to unequal sample sizes, a 1-sided Fisher's exact test was used to test the hypothesis that proportions of greater than or equal to 4-fold rises were higher in the vaccinated than in the placebo group. Statistical significance level was 0.05
Statistical Analysis 5: Comparison: RSV 276 Vaccine vs Placebo; Test type: Superiority; p < 0.01, Fisher Exact — [p-value comment as in outcome 7, analysis 4]

8. Primary Outcome: Serum RSV-neutralizing Antibody Titers
Description: Serum RSV-neutralizing antibody titers were assessed by 60% RSV-plaque reduction neutralization titer (RSV-PRNT) assay.
Time Frame: Measured at Day 56
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: log 2 titers
Arm/Group | RSV ΔNS2/Δ1313/I1314L Vaccine | RSV 276 Vaccine | Placebo
Number analyzed (Participants) | 25 | 24 | 12
log 2 titers | 5.1 [4.1 to 6.2] | 6.7 [6.0 to 7.8] | 2.3 [2.3 to 2.3]
Statistical Analysis 1: Comparison: RSV ΔNS2/Δ1313/I1314L Vaccine vs Placebo; Test type: Superiority; p < 0.01, Wilcoxon (Mann-Whitney) — Due to unequal sample sizes, a 1-sided Wilcoxon test was used to test the hypothesis that antibody levels at Day 56 were higher in the vaccinated than in the placebo group. Statistical significance level was 0.05
Statistical Analysis 2: Comparison: RSV 276 Vaccine vs Placebo; Test type: Superiority; p < 0.01, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 8, analysis 1]

9. Primary Outcome: Number of Participants With a Greater Than or Equal to 4-fold Rise in Serum Antibody Titers to RSV F Glycoprotein
Description: Antibodies were assessed by Enzyme-linked Immunosorbent Assay (ELISA). A response was defined as a greater than or equal to 4-fold increase in titer in paired specimens, between pre-inoculation and post-inoculation time points.
Time Frame: Measured at Day 0 and Day 56
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | RSV ΔNS2/Δ1313/I1314L Vaccine | RSV 276 Vaccine | Placebo
Number analyzed (Participants) | 25 | 24 | 12
Participants | 15 | 22 | 0
Statistical Analysis 1: Comparison: RSV ΔNS2/Δ1313/I1314L Vaccine; Test type: Other; % with >=4 fold rise in RSV F protein = 60, 90% CI 2-sided [42 to 76]
Statistical Analysis 2: Comparison: RSV 276 Vaccine; Test type: Other; % with >=4 fold rise in RSV F protein = 92, 90% CI 2-sided [76 to 98]
Statistical Analysis 3: Comparison: Placebo; Test type: Other; % with >=4 fold rise in RSV F protein = 0, 90% CI 2-sided [0 to 22]
Statistical Analysis 4: Comparison: RSV ΔNS2/Δ1313/I1314L Vaccine vs Placebo; Test type: Superiority; p < 0.01, Fisher Exact — [p-value comment as in outcome 7, analysis 4]
Statistical Analysis 5: Comparison: RSV 276 Vaccine vs Placebo; Test type: Superiority; p < 0.01, Fisher Exact — [p-value comment as in outcome 7, analysis 4]

10. Primary Outcome: Serum Antibody Responses to RSV F Glycoprotein
Description: Serum antibody titers to RSV F glycoprotein were assessed by ELISA.
Time Frame: Measured at Day 56
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: log 2 titers
Arm/Group | RSV ΔNS2/Δ1313/I1314L Vaccine | RSV 276 Vaccine | Placebo
Number analyzed (Participants) | 25 | 24 | 12
log 2 titers | 10.4 [9.3 to 11.8] | 12.6 [11.3 to 13.3] | 6.4 [4.6 to 7.9]
Statistical Analysis 1: Comparison: RSV ΔNS2/Δ1313/I1314L Vaccine vs Placebo; Test type: Superiority; p < 0.01, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 8, analysis 1]
Statistical Analysis 2: Comparison: RSV 276 Vaccine vs Placebo; Test type: Superiority; p < 0.01, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 8, analysis 1]

11. Secondary Outcome: Number of Participants Who Had RSV-associated Symptomatic, Medically Attended Respiratory and Febrile Illness, by Grade, Among Those Who Experienced Natural Infection With wt RSV During the Subsequent RSV Season
Description: The number of participants who had RSV-associated, symptomatic, medically attended respiratory and febrile illness (MAARI) among those who had indicators of natural infection with wt RSV were presented. Natural infection with wt RSV during the RSV season surveillance was defined as having either RSV detected in nasal washes collected during illness visits for MAARI events or a > 4-fold rise in serum antibodies from pre- to post-RSV season in the absence of RSV-associated medical events. A participant was only counted once in each MAARI category, and that was in the line corresponding to the highest grade adverse event they had in that category. These events were graded (Grade 1-mild to Grade 4-life-threatening) following protocol-defined grading system outlined in Table 5 and Table 6 in the protocol document.
Time Frame: Measured through participant's last study visit, up to a total of 6 to 10 months depending on when participants enrolled in the study
Population: Only participants who had RSV detected in nasal washes or had greater than or equal to 4 fold rise in serum antibodies from pre- to post-RSV season in the absence of RSV-associated medical events were included.
Measure: Count of Participants; unit: Participants
Arm/Group | RSV ΔNS2/Δ1313/I1314L Vaccine | RSV 276 Vaccine | Placebo
Number analyzed (Participants) | 11 | 5 | 4
Participants
  Medically Attended Fever: No adverse event | 9 | 4 | 4
  Medically Attended Fever: Grade 1 | 1 | 0 | 0
  Medically Attended Fever: Grade 2 | 1 | 0 | 0
  Medically Attended Fever: Grade 3 | 0 | 1 | 0
  Medically Attended Fever: Grade 4 | 0 | 0 | 0
  Medically Attended Otitis Media: No adverse event | 9 | 4 | 3
  Medically Attended Otitis Media: Grade 1 | 0 | 0 | 0
  Medically Attended Otitis Media: Grade 2 | 2 | 1 | 1
  Medically Attended Otitis Media: Grade 3 | 0 | 0 | 0
  Medically Attended Otitis Media: Grade 4 | 0 | 0 | 0
  Medically Attended URI: No adverse event | 9 | 2 | 3
  Medically Attended URI: Grade 1 | 0 | 0 | 0
  Medically Attended URI: Grade 2 | 2 | 3 | 1
  Medically Attended URI: Grade 3 | 0 | 0 | 0
  Medically Attended URI: Grade 4 | 0 | 0 | 0
  Medically Attended LRI: No adverse event | 10 | 3 | 3
  Medically Attended LRI: Grade 1 | 0 | 0 | 0
  Medically Attended LRI: Grade 2 | 1 | 2 | 1
  Medically Attended LRI: Grade 3 | 0 | 0 | 0
  Medically Attended LRI: Grade 4 | 0 | 0 | 0

12. Secondary Outcome: Magnitude of Serum RSV-neutralizing Antibody Responses in the Vaccine and Placebo Recipients Who Experienced Natural Infection With wt RSV During the Subsequent RSV Season.
Description: Only participants who had RSV detected in nasal washes or a greater than or equal to 4-fold rise in serum antibodies during the subsequent RSV season were included. RSV-neutralizing antibody titers were measured pre- and post-RSV surveillance season subsequent to the time of the inoculation.
Time Frame: as for outcome 11
Population: Only participants who had RSV detected in nasal washes or a greater than or equal to 4-fold rise in serum antibodies during the subsequent RSV season were included. One child from a set of twins was randomly selected and excluded from the analysis.
Measure: Median (Inter-Quartile Range); unit: log 2 titers
Arm/Group | RSV ΔNS2/Δ1313/I1314L Vaccine | RSV 276 Vaccine | Placebo
Number analyzed (Participants) | 11 | 4 | 4
log 2 titers
  Pre-RSV surveillance | 4.0 [2.3 to 6.6] | 6.1 [5.8 to 7.3] | 2.3 [2.3 to 2.3]
  Post-RSV surveillance | 10.1 [7.7 to 10.8] | 10.6 [8.0 to 11.3] | 5.9 [4.5 to 6.3]

ADVERSE EVENTS:
Time Frame: From study entry to end of study. The duration of follow-up for a given participant was between 6 and 10 months depending on time of enrollment.
Description: From day 0-28, all SAEs, solicited AEs, and unsolicited AEs, with the exception of the following if not treated with prescription medication or over the counter medications with antipyretic properties: diaper rashes, teething pain, and spitting up. SAEs and LRIs were reported according to DAIDS EAE Manual V2.0 (see References). From day 29-56, SAEs were collected. After day 56, from November 1 - March 31 of the following year, medically attended fever, LRI, URI and otitis media were collected.
Groups:
- RSV Delta NS2: Participants received a single dose of the RSV ΔNS2/Δ1313/I1314L vaccine at study entry (Day 0).
  RSV ΔNS2/Δ1313/I1314L: 10^6 plaque-forming units (PFU); administered as nose drops
- RSV 276: Participants received a single dose of the RSV 276 vaccine at study entry (Day 0).
  RSV 276: 10^5 PFU; administered as nose drops
- Placebo: Participants received a single dose of placebo at study entry (Day 0). Placebo: Isotonic diluent, administered as nose drops
Arm/Group | RSV Delta NS2 | RSV 276 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25 | 0/12
Serious Adverse Events (participants affected / at risk) | 1/25 | 0/25 | 0/12
Other Adverse Events (participants affected / at risk) | 21/25 | 21/25 | 8/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RSV Delta NS2 (N=25) | RSV 276 (N=25) | Placebo (N=12)
Mental status changes (Psychiatric disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RSV Delta NS2 (N=25) | RSV 276 (N=25) | Placebo (N=12)
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 1
Tympanic membrane disorder (Ear and labyrinth disorders) | 0 | 0 | 2
Tympanic membrane hyperaemia (Ear and labyrinth disorders) | 0 | 2 | 2
Eye discharge (Eye disorders) | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 1
Frequent bowel movements (Gastrointestinal disorders) | 0 | 1 | 1
Infantile vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Teething (Gastrointestinal disorders) | 2 | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 3 | 0
Pyrexia (General disorders) | 9 | 8 | 2
Bronchiolitis (Infections and infestations) | 0 | 0 | 1
Otitis externa (Infections and infestations) | 0 | 0 | 1
Otitis media acute (Infections and infestations) | 3 | 7 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 1
Purulent discharge (Infections and infestations) | 0 | 1 | 1
Respiratory syncytial virus infection (Infections and infestations) | 0 | 2 | 0
Sinusitis bacterial (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 4 | 2 | 2
Viral rash (Infections and infestations) | 0 | 2 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 4 | 1
Foreign body in ear (Injury, poisoning and procedural complications) | 0 | 0 | 1
Breath sounds abnormal (Investigations) | 0 | 0 | 1
Infant irritability (Nervous system disorders) | 0 | 0 | 1
Irritability (Psychiatric disorders) | 1 | 4 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 15 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 6 | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 16 | 19 | 6
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 0
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-06-10): https://cdn.clinicaltrials.gov/large-docs/29/NCT03227029/Prot_002.pdf
  • Statistical Analysis Plan (2020-09-09): https://cdn.clinicaltrials.gov/large-docs/29/NCT03227029/SAP_003.pdf
  • Informed Consent Form (2017-06-15): https://cdn.clinicaltrials.gov/large-docs/29/NCT03227029/ICF_000.pdf